CLINICAL TRIAL: NCT04702867
Title: Association Between Periodontal Bone Loss and Maxillary Sinus Changes Determined Using Cone Beam Computed Tomography - A Retrospective Study
Brief Title: Association Between Periodontal Bone Loss and Maxillary Sinus Changes.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Harshapopli27
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Maxillary Sinus Disease; Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontal bone loss group: The cases with level of alveolar crest more than 2 mm from the CEJ as measured using CBCT scan on mesial and distal sides of all premolar and molar teeth.
- Healthy group: The cases with level of alveolar crest equal to or less than 2 mm from the CEJ as measured using CBCT scan on mesial and distal sides of all premolar and molar teeth.

SUMMARY:
AIM AND OBJECTIVES:

AIM To determine the association between periodontal bone loss and maxillary sinus changes through cone beam computed tomography.

OBJECTIVES Primary objectives- 1. To compare the presence of maxillary sinus changes in patients with radiographic evidence of periodontal bone loss with healthy controls.

Secondary objectives-

1. To determine the correlation between severity of periodontal bone loss with the changes in maxillary sinus.
2. To compare the mean maxillary sinus mucosal thickening in patients with radiographic evidence of periodontal disease with healthy controls.

MATERIALS AND METHODOLOGY:

STUDY DESIGN A retrospective study will be conducted in the department of Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.

STUDY SETTING Hospital based study - CBCT volumes which are available in the archives of Oral Medicine and Radiology department will be evaluated.

STUDY PERIOD This study will be completed in 6 months. STUDY SUBJECTS CBCT volumes of patients who have undergone CBCT examination between May 2019 and December 2020 for various dental purposes will be evaluated and the volumes fulfilling the inclusion criteria will be included in the study. The subjects will be divided into 2 groups- Periodontal disease group and Healthy group, INCLUSION CRITERIA

1. Good quality images with visualization of maxillary sinus and maxillary posterior teeth of at least one side.

EXCLUSION CRITERIA

1. Signs of endodontic pathology like periapical radiolucency, root canal fillings etc.
2. Presence of metal artifacts interfering with the view of the maxilla.
3. Presence of trauma or pathologies such as tumours, cysts or malignancies that obscure the view of the region of interest.

SAMPLE SIZE A minimum sample size of 71 maxillary scans in each group has been calculated to expect a difference of 26.84% in the prevalence of the 2 groups as ascertained from a pilot study, at a significance level of 0.05 and a power of 90%.

Since group one will further be divided into 3 classes, a sample size of 225 in each group shall be taken.

METHODOLOGY

* CBCT volumes of patients who have undergone CBCT for various dental purposes between May 2019 to December 2020 available in the archives of Department of Oral medicine and radiology will be evaluated.
* These scans will be screened for radiographic evidence of periodontal disease i.e. horizontal or vertical bone loss and bone loss at the furcation.
* Further, the periodontal bone loss scans i.e. 225 will be divided into 3 groups of 75 each: mild (<25%), moderate (25-50%) and severe (>50%) according to the amount of bone loss.
* The group with no bone loss will be taken as the control group i.e. 225.
* Maxillary sinuses will be evaluated according to the following criteria; score range from 0 to 6 ; 0 - no mucosal changes.,1 - area without cortical bone and with soft tissue density, thickness >3 mm, parallel to sinus bone wall,2- sinus polyp, 3-antral pseudo cyst, 4- non-specific opacification,5- periostitis,6- antrolith.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data will be tabulated in Microsoft Excel sheet. The results will be expressed as the frequency (%) of maxillary and Mean + Standard deviation (SD) for maxillary sinus mucosal thickening. Normality of data will be assessed and Chi-square or student T test shall be used for non-parametric and parametric data respectively. All analysis will be performed by SPSS software version 21. A p value less than 0.05 will be considered significant for all outcomes.

DETAILED DESCRIPTION:
TITLE: "Association between Periodontal bone loss and Maxillary sinus changes determined using Cone beam computed tomography-A retrospective study." RATIONALE: Odontogenic maxillary sinusitis (OMS) is a type of inflammation of the maxillary sinus mucosa which results from dental infections such as chronic apical periodontitis, periodontal infections, tooth extractions and sinus lift procedures. The first and second molars are close to the floor of the maxillary sinus followed by the premolar teeth and occasionally canine.5In the otorhinolaryngological literature, the incidence of odontogenic sinusitis has been underreported in the past, with 10-12% of OMS cases attributed to odontogenic infections. However, recent studies are suggestive of a much higher incidence i.e. 40% of all cases of CMS.

Periodontal disease has been attributed as one of the causes of odontogenic maxillary sinusitis by various studies. The studies done so far offer some limitations such as lack of a control group, lack of corelation with disease severity, not taking focal sinus thickening adjacent to the infected tooth into consideration, small sample sizes and lack of clinical correlation.

Thus, this study aims to determine the association between periodontal disease and maxillary sinusitis through cone beam computed tomography in an Indian subpopulation attempting to overcome the limitations of the previous studies.

RESEARCH QUESTION P: Population (Patients with radiographic evidence of periodontal disease in their CBCT images) I: Intervention (none) C: Control(Patients with no evidence of periodontal disease in their CBCT images) O: Outcome (Radiographic signs of maxillary sinus changes) T: Time Frame (6 months) S: Study Design (Retrospective study) Setting in Haryana , India Is periodontal bone loss a risk factor for development of maxillary sinus changes?

AIM AND OBJECTIVES:

AIM To determine the association between periodontal bone loss and maxillary sinus changes through cone beam computed tomography.

OBJECTIVES Primary objectives- 1. To compare the presence of maxillary sinus changes in patients with radiographic evidence of periodontal bone loss with healthy controls.

Secondary objectives-

1. To determine the correlation between severity of periodontal bone loss with the changes in maxillary sinus.
2. To compare the mean maxillary sinus mucosal thickening in patients with radiographic evidence of periodontal disease with healthy controls.

MATERIALS AND METHODOLOGY:

STUDY DESIGN A retrospective study will be conducted in the department of Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.

STUDY SETTING Hospital based study - CBCT volumes which are available in the archives of Oral Medicine and Radiology department will be evaluated.

STUDY PERIOD This study will be completed in 6 months. STUDY SUBJECTS CBCT volumes of patients who have undergone CBCT examination between May 2019 and December 2020 for various dental purposes will be evaluated and the volumes fulfilling the inclusion criteria will be included in the study. The subjects will be divided into 2 groups- Periodontal disease group and Healthy group, INCLUSION CRITERIA

1. Good quality images with visualization of maxillary sinus and maxillary posterior teeth of at least one side.

EXCLUSION CRITERIA

1. Signs of endodontic pathology like periapical radiolucency, root canal fillings etc.
2. Presence of metal artifacts interfering with the view of the maxilla.
3. Presence of trauma or pathologies such as tumours, cysts or malignancies that obscure the view of the region of interest.

SAMPLE SIZE A minimum sample size of 71 maxillary scans in each group has been calculated to expect a difference of 26.84% in the prevalence of the 2 groups as ascertained from a pilot study, at a significance level of 0.05 and a power of 90%.

Since group one will further be divided into 3 classes, a sample size of 225 in each group shall be taken.

METHODOLOGY

* CBCT volumes of patients who have undergone CBCT for various dental purposes between May 2019 to December 2020 available in the archives of Department of Oral medicine and radiology will be evaluated.
* These scans will be screened for radiographic evidence of periodontal disease i.e. horizontal or vertical bone loss and bone loss at the furcation.
* Further, the periodontal bone loss scans i.e. 225 will be divided into 3 groups of 75 each: mild (<25%), moderate (25-50%) and severe (>50%) according to the amount of bone loss.
* The group with no bone loss will be taken as the control group i.e. 225.
* Maxillary sinuses will be evaluated according to the following criteria; score range from 0 to 6 ; 0 - no mucosal changes.,1 - area without cortical bone and with soft tissue density, thickness >3 mm, parallel to sinus bone wall,2- sinus polyp, 3-antral pseudo cyst, 4- non-specific opacification,5- periostitis,6- antrolith.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data will be tabulated in Microsoft Excel sheet. The results will be expressed as the frequency (%) of maxillary and Mean + Standard deviation (SD) for maxillary sinus mucosal thickening. Normality of data will be assessed and Chi-square or student T test shall be used for non-parametric and parametric data respectively. All analysis will be performed by SPSS software version 21. A p value less than 0.05 will be considered significant for all outcomes.

ETHICAL CONSIDERATION Ethical clearance will be obtained from the Bio-medical & Health Research Ethics Committee (BHRC), PGIDS Rohtak to conduct the study. Patient confidentiality would be maintained by not disclosing their details

ELIGIBILITY:
Inclusion Criteria:

* 1. Good quality images with visualization of maxillary sinus and maxillary posterior teeth of at least one side.

Exclusion Criteria:

- 1. Signs of endodontic pathology like periapical radiolucency, root canal fillings etc.

2. Presence of metal artifacts interfering with the view of the maxilla. 3. Presence of trauma or pathologies such as tumours, cysts or malignancies that obscure the view of the region of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CBCT volumes of patients who have undergone CBCT examination between May 2019 and December 2020 for various dental purposes will be evaluated and the volumes fulfilling the inclusion criteria will be included in the study. The subjects will be divided into 2 groups- Periodontal bone loss group and Healthy group
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the maxillary sinus. | 6 months
  * Maxillary sinuses will be evaluated according to the following criteria; score range from 0 to 6
  * 0 - no mucosal changes.
  * 1 - area without cortical bone and with soft tissue density, thickness >3 mm, parallel to sinus bone wall
  * 2- sinus polyp
  * 3-antral pseudo cyst
  * 4- non-specific opacification
  * 5- periostitis
  * 6- antrolith.
  * Maxillary sinuses will be evaluated according to the following criteria; score range from 0 to 6
  * 0 - no mucosal changes.
  * 1 - area without cortical bone and with soft tissue density, thickness >3 mm, parallel to sinus bone wall
  * 2- sinus polyp
  * 3-antral pseudo cyst
  * 4- non-specific opacification
  * 5- periostitis
  * 6- antrolith. USING CBCT VIEWER PROGRAM

SECONDARY OUTCOMES:
Thickness of mucosal lining of the maxillary sinus. | 6 months
  Measured using in built linear measurement tools in CBCT viewer program .

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India